CLINICAL TRIAL: NCT06772402
Title: An Open Label, Single Arm IIT Clinical Study Evaluating the Safety, Tolerability, and Preliminary Efficacy of GCB-001 in the Treatment of Patients With Delayed Onset Type 2 SMA Who Can Sit Alone But Cannot Walk.
Brief Title: GCB-001 in Treatment of Patients With Type II (SMA) Spinal Muscular Atrophy
Acronym: GITOPWTSMA
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Genecombio Ltd. (Other)
Collaborators: The Children's Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GCB-001-401
Record Dates: First submitted 2025-01-03; First posted 2025-01-13 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Spinal Muscular Atrophy Type 2
Keywords: Type II SMA; AAV; GCB-001
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental : Low dose (Experimental): Low dose is the first cohort of the study with a low dose level.
  Interventions: Genetic: GCB-001
- Experimental : High dose (Experimental): High dose is the first cohort of the study with a high dose level.
  Interventions: Genetic: GCB-001

INTERVENTIONS:
Genetic: GCB-001 — GCB-001 is a self-complementary AAV9 carrying a full length human SMN transgenetic product.

SUMMARY:
This study explored dose escalation of single-arm, open, single intrathecal injection in patients with delayed onset type 2 SMA. The investigator plans to conduct 2 cohorts. It is expected that each dose will be enrolled 3 subjects, with a total of 6 subjects aged from 2-12 years old.

For safety reasons, first subject of each dose cohort needs to complete a 30-day safety observation. After the researcher determines that the dosing is safe and tolerable, the next two subjects can be enrolled in the cohort; The follow-up dose cohort adopts a sentinel test design, with the first subject of each dose group being a sentinel.

During the DLT observation period, if the subject does not observe DLT and the researcher believes that continuing treatment can bring clinical benefits to the subject, the subject will continue to receive treatment; During the DLT observation period, if there is no occurrence of DLT or ≥ grade 2 adverse events related to the investigational drug, it will be escalated to the next dose. If the subject experiences grade ≥ 2 adverse events related to the study drug, the dose will be expanded to 3 subjects for further safety observation. Each subject in each dose cohort will be enrolled on a case by case basis.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 2 years and ≤ 12 years, gender not limited;
2. Meet the clinical diagnostic criteria for type 2 SMA, have an onset age form 6 months to 18 months, are diagnosed with SMN1 double allele pathogenic mutation, have 2-4 copies of SMN2 gene, and meet the clinical diagnostic criteria for SMA 5qSMA;
3. Capable of sitting alone but has never acquired the ability to walk independently (according to HFMSE standards, sitting alone: able to maintain a sitting position without hand support and count to 3 or more; walking independently: able to walk 4 or more steps without assistance);
4. The guardians of the subjects are able to understand and willing to comply with the requirements and procedures of protocol, voluntarily participate and sign the informed consent form.

Exclusion Criteria:

1. Researchers believe that gene replacement therapy may cause unnecessary risk of concomitant diseases, such as serious cardiovascular and cerebrovascular diseases, digestive tract diseases, liver and kidney dysfunction diseases, diabetes, known epilepsy, convulsions, convulsions or family history of psychosis;
2. Subjects who have participated in AAV gene therapy or have participated in or are currently participating in clinical trials of other SMA drugs;
3. Received treatment with Nordenafil Sodium Injection within 4 months prior to administration;
4. Received treatment with risperidone within 15 days prior to administration;
5. Subjects who have been treated with β 2 receptor agonists within 30 days prior to treatment (excluding inhaled salbutamol);
6. Subjects with allergic constitution, including those who are allergic or hypersensitive to prednisolone, other glucocorticoids or their excipients, and allergic to local anesthetics;
7. During the screening period, non-invasive ventilation support should be used for at least 12 hours per day;
8. The serum Anti-AAV9 neutralizing antibody titer is greater than 1:200.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
The rate of adverse events from baseline to 12 months after administration Assessed by CTCAE v4.0. | 0-12 months
AAV viral load after a single administration. | 0-12 months
  Detect the AAV viral load by central lab.
AAV viral immunogenicity after a single administration. | 0-12 months
  Detect the AAV viral immunogenicity by central lab.
AAV viral shedding after a single administration. | 0-12 months
  Detect the AAV viral shedding by central lab.
The change in total HFMSE (Hammersmith Functional Motor Scale Expanded) score from baseline at 12 months after a single administration | 0-12 months
  This 66-point scale (66 = very much improved, 0 = very much worse, etc.) is used by the clinician to assess the participant's performance status; higher scores indicate better status.
The change in total RULM (Revised Upper Limb Module) score from baseline at 12 months after a single administration | 0-12 months
  This 38-point scale (38 = very much improved, 0 = very much worse, etc.) is used by the clinician to assess the participant's performance status of upper limb; higher scores indicate better status.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital ZheJiang Univisity School Of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No